CLINICAL TRIAL: NCT00915330
Title: Transbronchial Needle Aspiration With and Without Rapid On-site Cytopathologic Evaluation in the Diagnostic Approach to Hilar/Mediastinal Adenopathy: A Randomized Controlled Trial.
Brief Title: Rapid On-site Cytopathologic Evaluation in the Diagnosis of Hilar/Mediastinal Adenopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Marco Patelli, Maggiore Bellaria Hospital
Allocation: Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-Trisolini
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Lung Cancer; Sarcoidosis; Tuberculosis
Keywords: Transbronchial needle aspiration; Bronchoscopy; Rapid on-site cytopathologic evaluation; Mediastinal lymphadenopathy; Hilar Lymphadenopathy
MeSH Terms: conditions — Lung Neoplasms; Sarcoidosis; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBNA alone (Active Comparator): Arm A: TBNA alone.
  Interventions: Procedure: TBNA
- TBNA with ROSE (Experimental): Arm B: TBNA with ROSE.
  Interventions: Procedure: Rapid on-site cytopathologic evaluation (ROSE); Procedure: TBNA

INTERVENTIONS:
Procedure: Rapid on-site cytopathologic evaluation (ROSE) — ROSE: examination in the endoscopy suite, by a pathologist, during the bronchoscopic procedure, of samples obtained with transbronchial needle aspiration.
  Arms: TBNA with ROSE
Procedure: TBNA — transbronchial needle aspiration

SUMMARY:
The purpose of this study is to determine whether rapid on-site cytopathologic evaluation (ROSE) can increase the diagnostic yield of transbronchial needle aspiration (TBNA) in the diagnosis of hilar and mediastinal lymphadenopathy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Hilar and/or mediastinal lymphadenopathy (> 1 cm on the short axis, as assessed by contrast-enhanced CT scan (computed tomography))

Exclusion Criteria:

* Uncontrolled coagulopathy
* Refusal to sign informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Examine the diagnostic yield of the TBNA with ROSE arm versus the diagnostic yield of TBNA alone arm | 6-12 months

SECONDARY OUTCOMES:
Examine the percentage of inadequate samples in the TBNA with ROSE arm versus the TBNA alone arm | 6-12 months
Examine the number of biopsy sites in the TBNA with ROSE arm versus the TBNA alone arm | 6-12 months
Examine the complication rate of bronchoscopy in the TBNA with ROSE arm versus the TBNA alone arm | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Patelli, MD, Principal Investigator — Maggiore Hospital
Locations (1):
- Maggiore Hospital, Bologna, Italy

REFERENCES:
- [Result] Diacon AH, Schuurmans MM, Theron J, Louw M, Wright CA, Brundyn K, Bolliger CT. Utility of rapid on-site evaluation of transbronchial needle aspirates. Respiration. 2005 Mar-Apr;72(2):182-8. doi: 10.1159/000084050. PMID 15824529
- [Result] Davenport RD. Rapid on-site evaluation of transbronchial aspirates. Chest. 1990 Jul;98(1):59-61. doi: 10.1378/chest.98.1.59. PMID 2361413
- [Result] Baram D, Garcia RB, Richman PS. Impact of rapid on-site cytologic evaluation during transbronchial needle aspiration. Chest. 2005 Aug;128(2):869-75. doi: 10.1378/chest.128.2.869. PMID 16100180
- [Result] Diette GB, White P Jr, Terry P, Jenckes M, Rosenthal D, Rubin HR. Utility of on-site cytopathology assessment for bronchoscopic evaluation of lung masses and adenopathy. Chest. 2000 Apr;117(4):1186-90. doi: 10.1378/chest.117.4.1186. PMID 10767258
- [Derived] Trisolini R, Cancellieri A, Tinelli C, Paioli D, Scudeller L, Casadei GP, Forti Parri S, Livi V, Bondi A, Boaron M, Patelli M. Rapid on-site evaluation of transbronchial aspirates in the diagnosis of hilar and mediastinal adenopathy: a randomized trial. Chest. 2011 Feb;139(2):395-401. doi: 10.1378/chest.10-1521. Epub 2010 Oct 28. PMID 21030491